CLINICAL TRIAL: NCT05436028
Title: TRIal to Evaluate TraNsvenous TrIcuspid Valve ReplacemenT With LuX-Valve Plus System in Patients With Severe or Greater Tricuspid Regurgitation -- SafetY and Clinical Performance
Brief Title: A Study to Evaluate the Safety and Performance of LuX-Valve Plus System for Tricuspid Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jenscare Scientific (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JSNL-CIP-TVS02-01CE
Record Dates: First submitted 2022-06-08; First posted 2022-06-28 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Tricuspid Regurgitation
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LuX-Valve Plus transvenous tricuspid valve and delivery system（LuX-Valve Plus System） (Experimental): The LuX-Valve Plus System is intended for the treatment of patients with at least severe TR who are determined by a Heart Team to be at high risk of traditional open-heart surgery.
  Interventions: Device: Transcatheter Tricuspid Valve Intervention

INTERVENTIONS:
Device: Transcatheter Tricuspid Valve Intervention — Due to unsustainable effect of medical therapy and high risks of surgical treatment, transcatheter tricuspid valve intervention (TTVI) has been a major field of study in the world in the last 10 years. TTVI could potentially reduce TR with lower periprocedural risk and improve the patient's clinical status and prognosis. Per the ESC guidelines for surgical and interventional treatment of tricuspid regurgitation (2021 ESC/EACTS Guidelines for the Management of Valvular Heart Disease), Transcatheter intervention for symptomatic secondary severe TR may be considered in inoperable patients at a Heart Valve Centre with expertise in the treatment of tricuspid valve disease (Class IIb).
  Transcatheter tricuspid treatment options can be divided into categories based on their mechanism of action: coaptation enhancement (edge-to-edge repair and spacer device), annuloplasty devices, caval valve implantation and valve replacement.

SUMMARY:
This is a prospective, single-arm, multi-center trial to evaluate the LuX-Valve Plus system for treating symptomatic at least severe TR in patients who are deemed high risk for tricuspid surgery.

Treatment with the LuX-Valve Plus system may enable patients with tricuspid regurgitation to have a complete tricuspid valve replacement with a minimally invasive approach.

Up to 150 subjects will be implanted at up to 24 institutions worldwide. No single institution will be allowed to register more than 25% of total subjects. There is no minimum number of subjects to be registered at any site.

Up to3 per site, may be implanted by operators without prior experience using the LuX-Valve Plus device to gain hands-on experience.Each site has a maximum of 3 roll-in cases. The data of roll-in subjects will not count towards the overall enrollment cap. Safety and performance results of roll-in subjects will be analyzed in subgroups.

All subjects will be evaluated at baseline, procedure, discharge, 30 days, 6 months, 1 year, 2 years, 3 years, 4 years, and 5 years post-procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥50 years at time of consent
2. Severe or greater TR (≥3+) assessed on transthoracic echocardiography by Echo Core Lab (ECL) using a 5-grade classification
3. New York Heart Association (NYHA) Class II-IV
4. In the judgment of the Site Heart Team, the subject has been adequately treated per applicable standards, including optimal medical therapy with diuretics
5. The Site Heart Team concur the benefit-risk analysis supports transcatheter tricuspid valve replacement per current guidelines for the management of valvular heart disease, and the subject is at high risk for tricuspid valve surgery.
6. Patient must be able to fully understand all aspects of the investigation that are relevant to the decision to participate, and provide a written informed consent
7. In France, patient is affiliated to a health social security regimen or equivalent

Exclusion Criteria:

1. Pulmonary arterial systolic pressure (PASP) > 60 mmHg by echo Doppler (unless right heart catheterization [RHC] demonstrates PASP ≤60 mmHg) or R heart catheterization OR PASP > 2/3 systemic BP with PVR > 5 Wood units after vasodilator challenge, in the absence of symptomatic hypotension or systolic BP < 90 mmHg.
2. Left Ventricular Ejection Fraction (LVEF) <35%
3. Evidence of intracardiac mass, thrombus or vegetation
4. Anatomical structures precluding proper device deployment or device vascular access, evaluated by echo or CT
5. Ebstein Anomaly or congenital right ventricular dysplasia
6. Surgical correction is indicated for other concomitant valvular disease (e.g., severe aortic, mitral and/or pulmonic valve stenosis and/or regurgitation) Subjects with concomitant valvular disease may treat their respective valve first, and wait 2 months before being reassessed for the trial.
7. Patients with valve prostheses implanted in the tricuspid valve
8. Pre-existing prosthetic valve(s) (other than tricuspid ones) with clinically significant prosthetic dysfunction
9. Sepsis or active endocarditis within 3 months, or infections requiring antibiotic therapy within 2 weeks prior to the planned procedure
10. Untreated clinically significant coronary artery disease requiring revascularization
11. Acute myocardial infarction or unstable ischemia-related angina within 30 days prior to the planned procedure
12. Any percutaneous coronary, intracardiac or carotid intervention within 30 days prior to the planned procedure
13. Cerebrovascular stroke (ischemic or bleeding) within prior 3 months to enrollment
14. Active peptic ulcer or active gastrointestinal (GI) bleeding within prior 3 months to enrollment
15. Inability to tolerate anticoagulation or antiplatelet therapy
16. Cardiogenic shock manifested by low cardiac output, vasopressor dependence, or mechanical hemodynamic support
17. Renal insufficiency (eGFR < 30 ml/min per the Cockcroft-Gault formula) and/or renal replacement therapy at the time of screening
18. Chronic liver failure or cirrhosis with MELD-Albumin Score ≥ 12
19. Severe lung disease or patient dependent on home oxygen and deemed unsuitable by the local heart team or eligibility committee for the study.
20. Futility with estimated life expectancy<12 months.
21. Subjects currently participating in another clinical trial of an investigational drug or device that has not yet completed its primary endpoint.
22. Pregnant or lactating; or female of childbearing potential with a positive pregnancy test within 14 days prior to intervention (contraceptive requirement is shown in Appendix XI)
23. Allergic to one or more of the substances contained in the implant and/or delivery system, including nitinol, tantalum, PET, PTFE, bovine pericardium, Pebax, PA, Polyurethane, Stainless steel.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2023-05-23 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
A composite endpoint of Major Adverse Event (MAE) at 30 days post procedure | 30 days post procedure
  A composite endpoint of Major Adverse Event (MAE) at 30 days post procedure, as listed below:
  Cardiovascular Mortality Myocardial Infarction (MI) Stroke New onset renal failure requiring unplanned dialysis or renal replacement therapy Severe Bleeding (includes fatal, life-threatening and extensive bleeding as defined by MVARC) Non-selective tricuspid valve surgery or transcatheter re-intervention post procedure Major cardiac structural complications Major access site and vascular complications Device-related pulmonary embolism New pacemaker implantation due to AV block

SECONDARY OUTCOMES:
Acute Secondary Endpoints-Device Success Rate | From the first skin incision for the investigational device to the time patient's exist from OR/Cath lab,assessed up to 24 hours post procedure.
  Device success is defined as successful deployment of the device and removal of the delivery system as planned, with no unplanned surgery related to the device or access procedure.
Acute Secondary Endpoints-Procedural Success Rate | 7-day post procedure, or at discharge if the subjects are discharged within 7 days after the procedure
  Device success without clinically significant PVL, as determined by the Echo Core Lab (ECL) assessment of a discharge TTE. Subjects who die or undergo tricuspid valve surgery before discharge are procedure failures.
Acute Secondary Endpoints-Clinical Success Rate at 30 days | at 30 days
  Procedural success without MAEs at 30 days.
Clinical and Functional Endpoints-All-cause mortality | at 30 days, 6 months, 12 months and annually until 5 years post-procedure
  All-cause mortality
Clinical and Functional Endpoints-Cardiovascular mortality | at 30 days, 6 months, 12 months and annually until 5 years post-procedure
  Cardiovascular mortality
Clinical and Functional Endpoints-Heart failure hospitalization | at 30 days, 6 months, 12 months and annually until 5 years post-procedure
  Heart failure hospitalization
Clinical and Functional Endpoints-Tricuspid valve surgery or transcatheter re-intervention | at 30 days, 6 months, 12 months and annually until 5 years post-procedure
  Tricuspid valve surgery or transcatheter re-intervention
Clinical and Functional Endpoints-NYHA Functional Class | at 30 days, 6 months, 12 months and annually until 5 years post-procedure
  NYHA Functional Class
Clinical and Functional Endpoints-Distance of 6-Minute Walk Test (6MWT) | at 30 days, 6 months, 12 months and annually until 5 years post-procedure
  Distance of 6-Minute Walk Test (6MWT)
Clinical and Functional Endpoints-Kansas City Cardiomyopathy Questionnaire (KCCQ) | at 30 days, 6 months, 12 months and annually until 5 years post-procedure
  Kansas City Cardiomyopathy Questionnaire (KCCQ)：Scores are transformed to a range of 0-100,in which higher scores reflect better health status.
Clinical and Functional Endpoints-Edema assessment | at 30 days, 6 months, 12 months and annually until 5 years post-procedure
  Edema assessment (1+ to 4+)
Echocardiographic Endpoints-TR Severity Grade | at baseline, 7-day post procedure, or at discharge if the subjects are discharged within 7 days after the procedure, 30 days, 6 months, 12 months and annually until 5 years post-procedure
  TR Severity Grade
Echocardiographic Endpoints-Vena Contracta Width | at baseline, 7-day post procedure, or at discharge if the subjects are discharged within 7 days after the procedure, 30 days, 6 months, 12 months and annually until 5 years post-procedure
  Vena Contracta Width
Echocardiographic Endpoints-Regurgitation Jet Area | at baseline, 7-day post procedure, or at discharge if the subjects are discharged within 7 days after the procedure, 30 days, 6 months, 12 months and annually until 5 years post-procedure
  Regurgitation Jet Area
Echocardiographic Endpoints-Effective Regurgitant Orifice Area (EROA) | at baseline, 7-day post procedure, or at discharge if the subjects are discharged within 7 days after the procedure, 30 days, 6 months, 12 months and annually until 5 years post-procedure
  Effective Regurgitant Orifice Area (EROA)
Echocardiographic Endpoints-Regurgitant Volume | at baseline, 7-day post procedure, or at discharge if the subjects are discharged within 7 days after the procedure, 30 days, 6 months, 12 months and annually until 5 years post-procedure
  Regurgitant Volume
Echocardiographic Endpoints-Mean Tricuspid valve inflow gradient | at baseline, 7-day post procedure, or at discharge if the subjects are discharged within 7 days after the procedure, 30 days, 6 months, 12 months and annually until 5 years post-procedure
  Mean Tricuspid valve inflow gradient
Echocardiographic Endpoints-Right Atrial Volume | at baseline, 7-day post procedure, or at discharge if the subjects are discharged within 7 days after the procedure, 30 days, 6 months, 12 months and annually until 5 years post-procedure
  Right Atrial Volume
Echocardiographic Endpoints-Right ventricular functions assessments:TAPSE | at baseline, 7-day post procedure, or at discharge if the subjects are discharged within 7 days after the procedure, 30 days, 6 months, 12 months and annually until 5 years post-procedure
  Right ventricular functions assessments:TAPSE
Echocardiographic Endpoints-Right ventricular functions assessments:fractional area change（FAC） | at baseline, 7-day post procedure, or at discharge if the subjects are discharged within 7 days after the procedure, 30 days, 6 months, 12 months and annually until 5 years post-procedure
  Right ventricular functions assessments:fractional area change（FAC）
Echocardiographic Endpoints-Right ventricular functions assessments:systolic tricuspid lateral annular tissue velocity S' | at baseline, 7-day post procedure, or at discharge if the subjects are discharged within 7 days after the procedure, 30 days, 6 months, 12 months and annually until 5 years post-procedure
  Right ventricular functions assessments:systolic tricuspid lateral annular tissue velocity S'
Echocardiographic Endpoints-Right ventricular functions assessments:Hepatic vein flow reversal | at baseline, 7-day post procedure, or at discharge if the subjects are discharged within 7 days after the procedure, 30 days, 6 months, 12 months and annually until 5 years post-procedure
  Right ventricular functions assessments:Hepatic vein flow reversal
Echocardiographic Endpoints-Right ventricular functions assessments:Inferior Cava Vein Diameter/respiratory variations | at baseline, 7-day post procedure, or at discharge if the subjects are discharged within 7 days after the procedure, 30 days, 6 months, 12 months and annually until 5 years post-procedure
  Right ventricular functions assessments:Inferior Cava Vein Diameter/respiratory variations
Echocardiographic Endpoints-Systolic pulmonary artery pressure | at baseline, 7-day post procedure, or at discharge if the subjects are discharged within 7 days after the procedure, 30 days, 6 months, 12 months and annually until 5 years post-procedure
  Systolic pulmonary artery pressure
Echocardiographic Endpoints-Cardiac Output | at baseline, 7-day post procedure, or at discharge if the subjects are discharged within 7 days after the procedure, 30 days, 6 months, 12 months and annually until 5 years post-procedure
  Cardiac Output
Echocardiographic Endpoints-Left Ventricular Ejection Fraction (LVEF) | at baseline, 7-day post procedure, or at discharge if the subjects are discharged within 7 days after the procedure, 30 days, 6 months, 12 months and annually until 5 years post-procedure
  Left Ventricular Ejection Fraction (LVEF)
Echocardiographic Endpoints-Paravalvular leak severity | at baseline, 7-day post procedure, or at discharge if the subjects are discharged within 7 days after the procedure, 30 days, 6 months, 12 months and annually until 5 years post-procedure
  Paravalvular leak severity

CONTACTS AND LOCATIONS:
Locations (1):
- Unité Médico-Chirurgicale, Hôpital Haut Lévêque, CHU de Bordeaux, Bordeaux, Gironde, France

IPD SHARING:
Plan to Share IPD: No